CLINICAL TRIAL: NCT02266901
Title: Transluminal or Percutaneous Endoscopic Drainage and Debridement of Abcesses After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Bariatric endoscopic drainage
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Obesity; Sepsis
Keywords: leaks after bariatric surgery; fistulae after bariatric surgery; abdominal abcesses and bariatric surgery; endoscopic drainage of abcesses; percutaneous drainage of abcesses; gastric bypass; sleeve gastrectomy; necrotic collection and bariatric surgery
MeSH Terms: conditions — Obesity; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cases (endoscopic drainage): Septic patients presenting post-bariatric collections related to leaks not adequately drained by percutaneous drain, for whom endoscopic drainage of the collections was performed by transluminal or percutaneous route.
  Interventions: Procedure: endoscopic drainage

INTERVENTIONS:
Procedure: endoscopic drainage — Endoscopic percutaneous access was obtained through surgical drains or after ultrasound-guided percutaneous drainage with a thin scope , and transluminal procedures with large scopes through the leak hole. All the procedures were performed under general anesthesia and carbon dioxide insufflation. Debridement was done by pus aspiration and irrigation.

SUMMARY:
Patients presenting intra-abdominal abcesses following bariatric surgery complicated by fistulae are classically treated by external drainage and endoprosthesis or surgical redo. Morbidity and mortality being increased in case of necrotic collections, an endoscopic debridement treatment might be proposed in certain cases. This present study aim to review the evolution of the patients treated by this method from 2007 to 2011 in the investigators institution.

DETAILED DESCRIPTION:
This retrospective study in an academic tertiary center will review the files of patients who underwent endoscopic drainage and debridement of abdominal abscesses secondary to bariatric surgery leaks . The decision for endoscopic treatment was made by the medico-surgical team in charge of this type of surgery, who had to weigh the high risk of mortality in case of re-intervention, along with endoscopic access to abscesses via the transluminal or percutaneous route based on abdominal imaging.

Data collection will lead to the evaluation of the technical success rate, the clinical success and potential complications.

ELIGIBILITY:
Inclusion Criteria:

* All the patient treated in an academic tertiary center who underwent endoscopic drainage and debridement of abdominal abscesses secondary to bariatric surgery leaks from october 2007 to April 2011
* septic state

Exclusion Criteria:

* All other necrosectomies performed for pancreatic disorders were excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All the patient treated in an academic tertiary center (Erasme Hospital) who underwent endoscopic drainage and debridement of abdominal abscesses secondary to postbariatric surgery leaks from october 2007 to April 2011. All other necrosectomies performed for pancreatic disorders were excluded from the study
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2007-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Intervention technical success | during the procedure
  success to pass the scope and perform abcess debridement of the targeted collection

SECONDARY OUTCOMES:
Clinical success | 7 days
  success to control sepsis after endoscopic drainage

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Devière, MD, PhD, Study Director — Erasme Hospital, ULB